CLINICAL TRIAL: NCT01629888
Title: A Clinical Study for Evaluating the Safety of Excessive Consumption of a Plant Sterol-enriched Yoghurt Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Japan (Industry)
Responsible Party: Sponsor
Organization: Danone Global Research & Innovation Center (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NU336
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Healthy; Mild Hypercholesterolemia
Keywords: Plant sterol; Hypercholesterolemia; dairy
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 = Tested product (Experimental)
  Interventions: Other: 1- plain low-fat dairy fermented product (drinkable) enriched with plant sterols-esters (1,6g /day equivalent as free sterols).
- 2 = Control product (Placebo Comparator)
  Interventions: Other: 2- plain low-fat dairy fermented product (drinkable) without plant sterols-esters

INTERVENTIONS:
Other: 1- plain low-fat dairy fermented product (drinkable) enriched with plant sterols-esters (1,6g /day equivalent as free sterols). — 1 = Intervention 1 (3 test products/day)
  Arms: 1 = Tested product
Other: 2- plain low-fat dairy fermented product (drinkable) without plant sterols-esters — 2 = Intervention 2 (3 control products/day)
  Arms: 2 = Control product

SUMMARY:
The purpose of this study is to investigate the safety of consumption of three times the standard dose of a yoghurt drink enriched with 1600 mg of plant sterols.

ELIGIBILITY:
Inclusion Criteria:

* male/female subjects,
* aged 20-65 years old,
* triglycerides (TG) levels under 400 mg/dL,
* total cholesterol plasma level under 240 mg/dL (with half the subjects at entry under 200 mg/dL),
* LDL-cholesterol plasma level under 160 mg/dL (with half the subjects at entry under 120 mg/dL),
* non diabetic and non hypertensive,
* accepting to follow the dietary recommendations advisable for hypercholesterolemic patient (Japan Atherosclerosis Society guidelines),
* effective contraceptive methods used for female subjects,
* having given written consent to take part in the study

Exclusion Criteria:

* subjects with sitosterolemia,
* subjects with 200 ml of blood taken within the past month or 400 ml or more within the past 3 months,
* taking any hypocholesterolemic treatment,
* presenting known allergy or hypersensitivity to plant sterols,
* dairy products and lactose, subject with heavy alcohol intake (> 60g/day),
* receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters,
* subjects receiving a transplant or under immunosuppressor treatment,
* receiving treatment for any serious pathology.
* for female subject:

  * pregnancy,
  * breast feeding or
  * intention to be pregnant during the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Senri Chuo Ekimae Clinic, Osaka, Japan